CLINICAL TRIAL: NCT06691971
Title: A Pilot Study to Assess Aevice Medical Device for Detection of Wheeze in Pediatric and Adult Populations
Brief Title: AeviceMD for Detection of Wheeze in Pediatric and Adult Populations
Status: Recruiting | Type: Observational
Sponsor: Aevice Health Pte. Ltd. (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: AE_MD_002
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-11

CONDITIONS: Subject Presenting Wheeze; Asthma; Bronchial Disease; Respiratory Tract Diseases; Pediatric Asthma; Chronic Respiratory Disease
Keywords: Wheeze; Auscultation; Wearable Medical Device
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients diagnosed with acute asthma exacerbation: Patients diagnosed with acute asthma exacerbation
  Interventions: Device: AeviceMD
- Patient with a non-cardiac AND non-pulmonary chief complaint and discharge diagnosis: Patient with a non-cardiac AND non-pulmonary chief complaint and discharge diagnosis

INTERVENTIONS:
Device: AeviceMD — The AeviceMD device will be placed on the patient to detect the presence of wheeze and perform auscultation.
  Other Names: AeviceMD Monitoring System
  Groups: Patients diagnosed with acute asthma exacerbation

SUMMARY:
Respiratory signs and symptoms consisting of wheeze, cough, and breathlessness are obtained in a manual fashion through history taking and physical examination by the healthcare professional. Auscultation of the lung assesses airflow through the trachea-bronchial tree and is helpful in diagnosing various respiratory disorders. AeviceMD is a wearable device that can acquire and process lung sounds, thus assisting in the detection of abnormal lung sounds. The primary objective of this study is to determine if AeviceMD can detect wheeze of pediatrics and adults as accurately as a physician through auscultation. The secondary objective is to investigate if AeviceMD can be used for remote auscultation of breath sounds.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and/or parents/guardians are able to give informed consent for participation in the study.
* Male or Female, aged ≥ 3 years.
* Diagnosed with acute asthma exacerbation by an ED provider.

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the subjects at risk because of participation in the study, or may influence the result of the study, or the subject's ability to participate in the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study will include 160 Subjects (80 Pediatrics and 80 Adult Subjects) who are presenting with wheeze in the emergency department, and outpatient and inpatient settings
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Wheeze is detected by physician and AeviceMD | 60 Seconds
  Primary endpoint of wheeze will be captured in a binary fashion (i.e. PRESENT or NOT PRESENT) on the CRF by the physician during manual auscultation. AeviceMD will perform wheeze analysis on each 5 sec of recording.

SECONDARY OUTCOMES:
Respiratory sounds are detected and identified by onsite physician and offsite (remote) physician | 150 Seconds
  Secondary endpoint of normal, abnormal and absent breath breath sounds will be captured in a binary fashion (i.e. PRESENT or NOT PRESENT) on the CRF by the physician during manual auscultation - i.e. bronchovesicular, crackles. Normal, abnormal and absent breath sounds will be annotated in a binary fashion (i.e. PRESENT or NOT PRESENT) on the CRF by the independent physician during remote auscultation - i.e. bronchovesicular, crackles.

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided